CLINICAL TRIAL: NCT02501837
Title: The Influence of Oxytocin on Pair-bonding and Emotion Regulation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Rene Hurlemann, Antragsteller und verantwortlicher Leiter, University Hospital, Bonn
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: OXT_BOND
Record Dates: First submitted 2015-07-15; First posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: Healthy women

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Experimental): 24 IU Oxytocin (Syntocinon spray), intranasal application 30 min prior to the experiment
  Interventions: Drug: Syntocinon-Spray
- Placebo (Placebo Comparator): Intranasal application, containing all ingredients except for the peptide, 3 puffs per nostril
  Interventions: Drug: Syntocinon-Spray

INTERVENTIONS:
Drug: Syntocinon-Spray — Intranasal administration of 24 IU Oxytocin

SUMMARY:
The neuropeptide oxytocin (OXT) has been identified as a key modulator of human social behavior and it has been recently shown that OXT also contributes to pair-bonding in men. However, it is still elusive whether OXT has similar effects in women. In the present study, the investigators examine the effect of intranasal OXT on behavioral ratings of and neural responses to the male partner in female participants. In a second experiment, the modulatory effect of OXT on emotion regulation is investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers
* In a heterosexual relationship

Exclusion Criteria:

* Current or past psychiatric disease
* Current or past physical illness
* Psychoactive medication
* Pregnant or lactating

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Neural response to photographs of the partner | About one hour after the intranasal administration of oxytocin
  Neural responses will be measured by using functional magnetic resonance imaging (fMRI). In the fMRI analysis the effect of oxytocin on the neural response to the photograph of the partner will be compared with placebo.
Neural response during the regulation of food craving | About one hour after the intranasal administration of oxytocin
  Neural responses will be measured by using functional magnetic resonance imaging (fMRI). In the fMRI analysis the effect of oxytocin on the neural response to the regulation of food craving will be compared with placebo.

SECONDARY OUTCOMES:
Attractiveness ratings of all stimuli | About one hour after the intranasal administration of oxytocin
  The effect of oxytocin on attractiveness ratings of the partner will be compared with placebo. Ratings will be obtained by using a visual analog scale.
Arousal ratings of all stimuli | About one hour after the intranasal administration of oxytocin
  The effect of oxytocin on arousal ratings of the partner will be compared with placebo. Ratings will be obtained by using a visual analog scale.
Food craving ratings | About one hour after the intranasal administration of oxytocin
  The effect of oxytocin on food craving ratings will be compared with placebo. Ratings will be obtained by using a visual analog scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, University of Bonn, Bonn, Germany

REFERENCES:
- See also: Homepage of the research group — http://renehurlemann.squarespace.com/welcome/